CLINICAL TRIAL: NCT05142553
Title: A Phase IIb, Double-blind, Randomised, Active-controlled, Multi-centre, Non-inferiority Trial Followed by a Phase III, Single-arm, Open-label Trial, to Assess Immunogenicity and Safety of a Booster Vaccination With a Recombinant Protein RBD Fusion Dimer Candidate (PHH-1V) Against the Virus That Cause COVID-19, Know as Severe Acute Respiratoy Syndrome Coronavirus 2 (SARS-CoV-2)SARS-CoV-2, in Adults Fully Vaccinated Against COVID-19 Followed by an Extension Period to Study a Fourth Dose Administration of PHH-1V.
Brief Title: Immunogenicity and Safety of a Booster Vaccination With a Recombinant Protein RBD Candidate Vaccine Against SARS-CoV-2 in Healthy Adults Volunteers Fully Vaccinated Followed by an Extension Period to Study a Fourth Dose Administration.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hipra Scientific, S.L.U (Industry)
Collaborators: Laboratorios Hipra, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HIPRA-HH-2
Record Dates: First submitted 2021-11-17; First posted 2021-12-02 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; SARS-CoV-2 Acute Respiratory Disease
MeSH Terms: conditions — COVID-19 | interventions — HIPRA COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: This is a Phase IIb, randomised, double-blind, active-controlled, multicentre, noninferiority clinical study that aims to determine immunogenicity, reactogenicity, safety, and tolerability of a booster vaccination of test vaccine followed by an extension period to study a fourth dose administration of the vaccine.
Who Masked: Participant, Investigator
Masking Description: Subjects and the clinical study team will remain blinded to treatment allocation. Clinical staff involved in study drug preparation and administration will be aware of which vaccine the subject is receiving. The extension of the fourth dose will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Vaccine HIPRA (Experimental): 40 ug/0.5 ml
  Interventions: Biological: COVID-19 Vaccine HIPRA
- Cominarty (Pfizer-BioNtech) (Active Comparator): 30 micrograms/dose concentrate for dispersion for injection
  Interventions: Biological: Cominarty (Pfizer-BioNtech)

INTERVENTIONS:
Biological: COVID-19 Vaccine HIPRA — Subjects will receive one injection of COVID-19 Vaccine HIPRA
  Arms: COVID-19 Vaccine HIPRA
Biological: Cominarty (Pfizer-BioNtech) — Subjects will receive one injection of Cominarty Vaccine
  Arms: Cominarty (Pfizer-BioNtech)

SUMMARY:
This Phase IIb clinical study aims to compare the immunogenicity and safety of a booster dose of recombinant protein RBD fusion dimer vaccine as a heterologous booster (to subjects who have received the second dose of the Pfizer-BioNTech (Comirnaty) COVID-19 vaccine at least 182 days prior to the booster dose in this study) versus a homologous booster (subjects who received the second dose of the Comirnaty COVID-19 vaccine at least 182 days prior to the booster dose in this study) will receive a third dose of the Comirnaty vaccine).

The extension part of the study aims to compare the immunogenicity and safety of a fourth dose of PHH-1V in subjects with a primovaccination with Pfizer-BioNTech (Comirnaty) COVID-19 vaccine plus either a booster dose of Comirnaty or PHH-1V versus those with three vaccinations of Comirnaty.

DETAILED DESCRIPTION:
The study population includes 1075 healthy adults aged above 18 years old who have received two doses of the Comirnaty vaccine, and are at least 182 days and less than 365 days after their second dose will be randomly assigned to two treatment arms. In each arm, volunteers will be randomized in a ratio Test vaccine:Comirnaty of 2:1. Each participant will receive one booster immunisation and will be followed for 1 year to evaluate immunogenicity response and assess the safety of the test vaccine in comparison to Cominarty.

The study population of the extension part includes 200 healthy adults abode 18 years old who have received or: 3 doses of Comirnaty vaccine, or 2 doses of Comirnaty + 1 dose of PHH-1V. Each participant will receive one dose of PHH-1V.

ELIGIBILITY:
Part A: Inclusion Criteria:

* Male or female, by birth, ≥ 18 years old at Screening.
* Willing and able to comply with scheduled visits, laboratory tests, complete diaries, and other study procedures.
* Body Mass Index (BMI) between 18 to 40 kg/m2.
* Has received a complete COVID-19 vaccination programme (two administrations, prime and boosting) at least 182 days and with a maximum of 365 days before Screening with Comirnaty vaccine.
* Has a negative COVID-19 polymerase chain reaction (PCR) test at Screening.
* Willing to avoid all other vaccines within 4 weeks before and after vaccination in this study (Day 0). Seasonal influenza vaccination is allowed if it is received at least 14 days before or after vaccination.
* Willing to refrain from blood donation during the study.
* Women of childbearing potential must have a negative urine pregnancy test at Screening and prior to vaccination.
* Women of childbearing potential must be willing to use highly effective contraceptive methods or have practiced sexual abstinence from the screening visit until 8 weeks after the vaccination.
* Males who are not sterilised, must be willing to avoid impregnating female partners from Screening until 8 weeks after vaccination.
* Willing and able to provide written informed consent prior the initiation of any study procedures.

Part A: Exclusion criteria:

* Pregnant or lactating or intending to become pregnant or plans to breastfeed during the study.
* Positive pregnancy test at Screening or vaccination day.
* Any medical disease (acute, subacute, intermittent, or chronic) or condition that in the opinion of the Investigator compromises the subject's safety, preclude vaccination or compromises interpretation of the results.
* Ongoing serious psychiatric condition likely to affect participation in the study (e.g., ongoing severe depression, recent suicidal ideation, bipolar disorder, personality disorder, alcohol and drug dependency, severe eating disorder, psychosis, use of mood stabilisers or antipsychotic medication).
* History of respiratory disease (e.g., chronic obstructive pulmonary disease [COPD]) requiring daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 6 months.
* History of significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult. Controlled hypertension will be permitted at the discretion of the Investigator.
* History of neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, or transverse myelitis).
* Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
* Any confirmed or suspected autoimmune, immunosuppressive or immunodeficiency disease/condition (iatrogenic or congenital), including human immunodeficiency virus (HIV) infection, asplenia, or recurrent severe infections.
* Acute illness within 72 hours before vaccination day that, in the opinion of the Investigator may interfere the evaluation of safety parameters.
* Received investigational drug within 90 days before Screening or plans to participate in another interventional clinical study (drug/biologic/device) within 12 months after vaccination.
* History of hypersensitivity or severe allergic reactions, including anaphylaxis, generalised urticarial, angioedema and other significant reactions related to food, drugs, vaccines, or pharmaceutical agents, which are likely to be exacerbated by any component of the COVID-19 vaccine HIPRA.
* Use of any immunosuppressant, glucocorticoids, or other immune-modifying drugs within 2 months before vaccination day; or anticipation of the need for immunosuppressive treatment within 182 days after vaccination.
* Received immunoglobulin, blood-derived products, or other immunosuppressant drugs within 90 days before vaccination (Day 0).
* Known disturbance of coagulation (iatrogenic or congenital) or blood dyscrasias.
* Known bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), (iatrogenic or congenital), blood dyscrasias, or prior history of significant bleeding or bruising following intramuscular (IM) injections or venepuncture.
* Chronic liver disease.
* Positive test for HIV types 1 or 2 infection, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies (HCV Abs) at Screening.
* Suspected or known current alcohol abuse or any other substances abuse (except tobacco).

History of COVID-19 infection.

* Ever been included in a trial with an experimental vaccine against COVID-19.
* Close contact with anyone known to have SARS-CoV-2 infection within 15 days before Screening.
* Scheduled elective surgery during the study.
* Life expectancy of less than 12 months.
* Any condition and/or laboratory finding that, in the Investigators opinion, would interfere with the study or put the subject at risk.

Part B (fourth dose extension): Inclusion Criteria

* Adults ≥ 18 years old at Day 0.
* Participant must provide consent indicating that she or he understands the purpose and potential risks and is willing and able to participate in this extension of the study and comply with all the study requirements and procedures.
* Has received a primary vaccination of two doses of Comirnaty followed by a booster dose either with Comirnaty or PHH-1V. Last booster dose given between 6 and 12 months before Day 0.
* Has a negative Rapid Antigen Test (RAT) at Day 0 before the fourth dose administration.
* Participants may have underlying illnesses if are stable and well-controlled.
* Participant is willing to avoid receiving live attenuated vaccines (licensed) within 4 weeks before screening or after receiving any study vaccine, or other not live vaccines (licensed) within 14 days before and after receiving any study vaccine.
* Participant agrees not to donate blood, blood products and bone marrow at least 12 weeks before and after vaccination
* Contraceptive use for women of childbearing potential: hormonal, intrauterine device, vasectomized partner, sexual abstinence, condom.
* Negative pregnancy test for WOCBP at Day 0.
* Contraceptive use for males: vasectomized participants, condom, sexual abstinence.

Part B (fourth dose extension): Exclusion Criteria

* History of anaphylactic shock of any kind
* History of COVID-19 infection.
* Pregnancy or breast-feeding at screening or Day 0
* Participant has a clinically significant acute illness or fever (temperature ≥38º C / 100.4ºF) at screening or within 48 hours prior to the planned vaccination
* Participant had a surgery requiring hospitalization before vaccination and he/she has not received the hospital discharge at day 0
* Participant has any active malignancy
* Participant has ongoing severe and non-stable psychiatric condition likely to affect participation in the study
* Participant has a problematic or risk use of substances including alcohol that can compromise the study follow-up
* Participant has a bleeding disorder, blood dyscrasia, or continuous use of anticoagulants or has any condition that contraindicates intramuscular injections or frequent phlebotomy
* Participant has abnormal function of the immune system as in autoimmune diseases, asplenia, recurrent infections or congenital/acquired immunodeficiency
* Chronic or recurrent administration (during at least 14 days) of systemic immunosuppressant medication within 12 weeks preceding the planned administration of study vaccine
* Subject has received immunoglobulins and/or blood-derived products 12 weeks prior vaccination
* Participant received any immunotherapy (monoclonal antibodies, plasma) aimed to prevent or treat COVID-19 within 90 days preceding the planned administration of study vaccine
* Participation in any research involving an investigational product (drug, biologic, device) within 12 weeks prior to vaccination and during the study
* Participant has donated ≥ 450ml of blood products within 12 weeks before screening
* Participant has any medical condition and/or finding that in the investigator opinion might increase participant risks, interfere with the study or impair interpretation of study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 887 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Part A: Changes of the immunogenicity against Wuhan | 14 days
  Neutralisation titre measured as inhibitory concentration 50 (IC50) for each individual sample and geometric mean titre (GMT) for treatment group comparison at Baseline and Day 14.
Safety and tolerability of PHH-1V as third or fourth dose | 7 days
  Number, percentage, and characteristics of solicited local reactions through Day 7 after vaccination.
Safety and tolerability of PHH-1V as third or fourth dose | 28 days
  Number, percentage, and characteristics of unsolicited local and systemic adverse events (AEs) through Day 28 after vaccination.
Safety and tolerability of PHH-1V as third or fourth dose | 364 days
  Number and percentage of serious adverse events (SAEs), adverse event of special interest (AESI) and medically attended adverse events (MAAE) through Day 364.
Safety and tolerability of PHH-1V as third or fourth dose | Days 14, 28, 182, and 364
  Change from baseline in safety laboratory parameters at Days 14, 28, 182, and 364 after vaccination.
Part B: Changes of the immunogenicity against Omicron BA.1 | Day 14
  Neutralisation titre measured as inhibitory concentration 50 (IC50) by PBNA and reported as log10 concentration for each individual sample and GMT, at Day 14 post-dose 4 of PHH-1V in cohort 2 versus post-dose 3 in cohort 2 (cohort 2 having three doses of Comirnaty + the frouth dose of PHH-1V).

SECONDARY OUTCOMES:
Changes of the immunogenicity against the Variants of Concern (VOC) | Day 14, 28, 98, 182, 364
  Neutralisation titre against VOC measured as IC50 for each individual sample and GMT for treatment group comparison at Baseline and Days 28, 98, 182, and/or 364.
Changes of the immunogenicity against the Variants of Concern (VOC) | Day 14, 28, 98, 182 and 364
  Geometric mean fold rise (GMFR) in neutralising antibodies titres for treatment group comparison at Baseline and Days 14, 28, 98, 182, and/or 364.
Changes of the immunogenicity against the Variants of Concern (VOC) | Day 14, 28, 98, 182 and 364
  Neutralisation titre against VOC measured as IC50 by PBNA and reported as reciprocal concentration for each individual sample and GMT for treatment group comparison at Baseline and Days 14, 28, 98, 182, and 364.
Changes of the immunogenicity against the Variants of Concern (VOC) | Day 14, 28, 98, 182 and 364
  Geometric mean fold rise (GMFR) in neutralising antibodies titres for treatment group comparison at Baseline and Days 14, 28, 98, 182, and 364.
Changes in immunogenicity at Baseline and Days 14, 28, 182 &364. | Days 14, 28, 98, 182 and 364
  Neutralisation titre measured as inhibitory dilution 50 (ID50) for each individual sample, and GMT for treatment group comparison at Baseline and Days 14, 28, 98, 182, and 364. This analysis will be performed in a subset of subjects.
Immunogenicity to the SARS-CoV-2 spike glycoprotein | Days 14, 28, 98, 182, and 364
  Percentage of subjects that, after a booster dose, have a ≥4-fold change in binding antibodies titre from Baseline and Days 14, 28, 98, 182, and 364.
T-cell mediated responses against the SARS-CoV-2 S glycoprotein at Baseline & D14. | Day 14
  T-cell-mediated response to the SARS-CoV-2 S protein at Baseline and at Day 14. This analysis will be performed in a subset of subjects.
Th-1/Th-2 T-cell mediated responses against the SARS-CoV-2 S glycoprotein at Baseline & D14. Th-1/Th2 | Day 14
  CD4+/CD8+ T-cell response to the SARS-CoV-2 S protein at Baseline and at Day 14. This analysis will be performed in a subset of subjects.

OTHER OUTCOMES:
Number of subjects with SARS-CoV-2 infections in subjects without evidence of infection before study's participation. | 364 Days
  Number and percentage of subjects with SARS-CoV-2 infections according to COVID-19 infection criteria throughout the study duration.
Number of COVID-19 severe infections after receiving PHH-1V. | through Day 364.
  Number and percentage of COVID 19 severe infections through Day 364.
Number of COVID-19 severe infections after receiving PHH-1V. | through Day 364.
  Number and percentage of hospital admissions associated with COVID 19 through Day 364.
Number of COVID-19 severe infections after receiving PHH-1V. | through Day 364.
  Number and percentage of intensive care unit (ICU) admissions associated with COVID-19 through Day 364.
Number of COVID-19 severe infections after receiving PHH-1V. | through Day 364.
  Number and percentage of deaths associated with COVID-19 through Day 364.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Prat, Study Chair — HIPRA SCIENTIFIC
Locations (10):
- Spain (10):
  - Hospital Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Principe de Asturias, Meco, Madrid
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Vall Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corominas J, Garriga C, Prenafeta A, Moros A, Canete M, Barreiro A, Gonzalez-Gonzalez L, Madrenas L, Guell I, Clotet B, Izquierdo-Useros N, Raich-Regue D, Gallemi M, Blanco J, Pradenas E, Trinite B, G Prado J, Perez-Caballero R, Bernad L, Plana M, Esteban I, Aurrecoechea E, Taleb RA, McSkimming P, Soriano A, Nava J, Anagua JO, Ramos R, Marti Lluch R, Corpes Comes A, Otero Romero S, Martinez-Gomez X, Camacho-Arteaga L, Molto J, Benet S, Bailon L, Arribas JR, Borobia AM, Queiruga Parada J, Navarro-Perez J, Forner Giner MJ, Lucas RO, Vazquez Jimenez MDM, Lopez Fernandez MJ, Alvarez-Mon M, Troncoso D, Arana-Arri E, Meijide S, Imaz-Ayo N, Garcia PM, de la Villa S, Rodriguez Fernandez S, Prat T, Torroella E, Ferrer L. Humoral and cellular immune responses after 6 months of a heterologous SARS-CoV-2 booster with the protein-based PHH-1V vaccine in a phase IIb trial. Vaccine. 2025 Feb 15;47:126685. doi: 10.1016/j.vaccine.2024.126685. Epub 2025 Jan 13. PMID 39809095
- [Derived] Moros A, Prenafeta A, Barreiro A, Perozo E, Fernandez A, Canete M, Gonzalez L, Garriga C, Pradenas E, Marfil S, Blanco J, Cebollada Rica P, Sistere-Oro M, Meyerhans A, Prat Cabanas T, March R, Ferrer L. Immunogenicity and safety in pigs of PHH-1V, a SARS-CoV-2 RBD fusion heterodimer vaccine candidate. Vaccine. 2023 Aug 7;41(35):5072-5078. doi: 10.1016/j.vaccine.2023.07.008. Epub 2023 Jul 16. PMID 37460353
- [Derived] Corominas J, Garriga C, Prenafeta A, Moros A, Canete M, Barreiro A, Gonzalez-Gonzalez L, Madrenas L, Guell I, Clotet B, Izquierdo-Useros N, Raich-Regue D, Gallemi M, Blanco J, Pradenas E, Trinite B, Prado JG, Blanch-Lombarte O, Perez-Caballero R, Plana M, Esteban I, Pastor-Quinones C, Nunez-Costa X, Taleb RA, McSkimming P, Soriano A, Nava J, Anagua JO, Ramos R, Lluch RM, Comes AC, Romero SO, Gomez XM, Sans-Pola C, Molto J, Benet S, Bailon L, Arribas JR, Borobia AM, Parada JQ, Navarro-Perez J, Forner Giner MJ, Lucas RO, Jimenez MDMV, Compan SO, Alvarez-Mon M, Troncoso D, Arana-Arri E, Meijide S, Imaz-Ayo N, Garcia PM, de la Villa Martinez S, Fernandez SR, Prat T, Torroella E, Ferrer L. Safety and immunogenicity of the protein-based PHH-1V compared to BNT162b2 as a heterologous SARS-CoV-2 booster vaccine in adults vaccinated against COVID-19: a multicentre, randomised, double-blind, non-inferiority phase IIb trial. Lancet Reg Health Eur. 2023 May;28:100613. doi: 10.1016/j.lanepe.2023.100613. Epub 2023 Apr 14. PMID 37131861